CLINICAL TRIAL: NCT06785610
Title: A Single-center, Single-arm Prospective Study to Evaluate Capsulase for Prevention of Capsular Contracture in Postmastectomy Patients Undergoing Implant-based Reconstructions
Brief Title: Prevention of Capsular Contracture in Postmastectomy Patients Undergoing Implant-based Reconstructions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UID 4634; L2-269 (Other: Comitato Etico Territoriale Lombardia 2)
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Capsular Contracture Associated With Implant
Keywords: Capsular Contracture; Mastectomy reconstruction; Definitive silicone implant

STUDY DESIGN:
Intervention Model Description: Single-center, single-arm prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capsulase® supplementation (Experimental): Capsulase® supplementation in the postoperative period
  Interventions: Dietary Supplement: Capsulase®

INTERVENTIONS:
Dietary Supplement: Capsulase® — Capsulase® supplement daily administration after surgery

SUMMARY:
The study plans to evaluate capsular contracture at 1-year follow-up in postmastectomy patients receiving immediate implant-based reconstruction and Capsulase® supplementation in the postoperative period. These data are compared with historical data of capsular contracture in patients not receiving any food supplementation postoperatively.

Aim of the study is to collect preliminary data to support Capsulase® supplementation in the postoperative period to prevent capsular contracture.

DETAILED DESCRIPTION:
Capsular contracture is one of the most common complications of breast implant use, in both reconstructive and aesthetic setting. Research on capsular contracture has focused on reducing bacterial contamination of implant surfaces through antibiotic and antiseptic solutions and, more recently, on the pharmacological control of the inflammation process around the implant. The foreign body reaction is responsible for capsular contracture.

Several experimental studies have demonstrated that it is possible to pharmacologically control the inflammation process around implants reducing the profibrotic substances included in the inflammation pathway.

Among diet supplements there are several substances that have been studied for their anti-inflammatory properties, in particular omega-3 fatty acids and boswellic acids.

Capsulase® is a diet supplement and consists of Boswellia serrata phospholipid INDENA®, palmitoylethanolamide (PEA), quercetin phytosome INDENA®, bromelain 2500 Gelatin Dissolving Units/gram (GDU/g) and vitamin E acetate. Its efficacy and safety in women with contracted breast implants have been evaluated both in the reconstructive and aesthetic setting. Although preliminary results are satisfactory, however the series include a small sample of women.

Aim of this study is to collect preliminary data to support Capsulase® supplementation in the postoperative period to prevent capsular contracture, comparing capsular contracture in postmastectomy patients receiving immediate implant-based reconstruction and Capsulase® supplementation in the postoperative period with historical data of capsular contracture in patients not receiving any food supplementation postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Immediate post mastectomy reconstruction with definitive silicone implant (microtextured prosthesis) (both therapeutic and risk reducing mastectomies)
* Informed consent
* Unilateral and bilateral mastectomies

Exclusion Criteria:

* Hypersensitivity to Capsulase®
* Pregnant women
* Impossibility of immediate reconstruction with definitive implants due to inadequacy of mastectomy flaps (inadequate in quantity and/or quality)
* Patients with previous breast implants
* Revisional surgery for capsular contracture
* Use of micro polyurethane foam-coated implants
* Mesh and matrix-assisted reconstructions
* Reconstruction of previous irradiated breasts

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Capsular contracture rate | 1 year
  Number of capsular contracture at 1-year follow-up

SECONDARY OUTCOMES:
Capsular contracture rate compared to historical data | 1 year
  Capsular contracture rate at 1-year in patients receiving Capsulase® supplementation compared with capsular contracture rate in the historical control arm of patients not receiving any supplementation
Patient satisfaction | 1 year
  Completion of BREAST-Q questionnaire (higher answers to each item reflect a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca De Lorenzi, MD, Principal Investigator — European Istitute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy